CLINICAL TRIAL: NCT05607342
Title: Pilot of Osanetant to Reduce Testosterone in Men With Adenocarcinoma of the Prostate (PORT-MAP)
Brief Title: Pilot of Osanetant to Reduce Testosterone in Men With Adenocarcinoma of the Prostate
Acronym: PORT-MAP
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Development of the drug program has been discontinued
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00148767
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — SR 142801

STUDY DESIGN:
Intervention Model Description: Single arm, pilot clinical trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pilot Trial: Osanetant 28 Days (Experimental): Pilot Trial: A single dose level (200mg twice daily, oral) will be provided for men with prostate cancer undergoing curative intent surgery. Men will undergo serum testing at baseline, days 2, 3, 7, 14, and 28 as well as 6 weeks post-treatment in order to evaluate efficacy. All men enrolled will be subject to the same study procedures and assessments, regardless of completion of the study protocol, and analysis will occur via intent-to-treat principles.
  Interventions: Drug: Osanetant

INTERVENTIONS:
Drug: Osanetant — To evaluate the effect of Osanetant on the testosterone levels.

SUMMARY:
To evaluate the effect of Osanetant on testosterone levels in men with prostate cancer within 28 days of therapy.

DETAILED DESCRIPTION:
Primary:

To evaluate the effect of Osanetant on testosterone levels in men with prostate cancer within 28 days of therapy.

Secondary:

* To evaluate the effect Osanetant on pituitary hormones (LH/FSH) and estrogen within 28 days of therapy.
* To evaluate the effect of Osanetant on PSA levels after 28 days (approximately 4 weeks) of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Males ≥ 18 years
* Histologic diagnosis of adenocarcinoma of the prostate (PCa)
* Planned radical prostatectomy within the study period
* Testosterone >150ng/ml
* Adequate organ function, defined as follows: Result Date

  * Leukocytes >1.5K/UL
  * Absolute Neutrophil Count >1.5K/UL
  * NOTE: Patients with established diagnosis of benign neutropenia are eligible to participate with ANC between 1000-1500 if in the opinion of treating physician the trial treatment does not pose excessive risk of infection to the patient.
* Platelets >100K/UL
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation
* Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
* Men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation. Men of child-bearing potential must not father a child or donate sperm while receiving investigational treatment. Following treatment (standard of care prostatectomy) there is no further child-bearing potential.

Exclusion Criteria:

* Current or recent (within 6 months) use of testosterone/estrogen modulating agents (leuprolide, degarelix, bicalutamide, enzalutamide, apalutamide, darolutamide, abiraterone, systemic ketoconazole, tamoxifen, etc)
* Current use of CYP3A4 inhibitors
* Subjects using the following medications within 2 weeks prior to first dosing (or within 5 times the half-life of that medication, whichever is longer) will be excluded from the study:

  * Inhibitors of CYP3A4 (including but not limited to macrolide antibiotics, HIV protease inhibitor, azole antifungal drugs, cyclosporine, calcium channel inhibitor, cimetidine)
  * Inducers of CYP3A4 (including but not limited to rifampicin, carbamazepine, efavirenz, bosentan, modafinil, St. John's Wort), Medications with narrow therapeutic index that are metabolized CYP3A4 and/or CYP2D6 are not allowed from screening until up to 5 half-lives after last dose of Osanetant is administered.
* Cognitive impairment (defined as the presence of diagnosed dementia)
* Impaired renal function: Cr >1.8
* Medical history of osteoporosis
* Current systemic corticosteroid, long-term opioid, spironolactone, or eplerenone use
* Has a known allergic reaction to any excipient contained in the study drug formulation
* Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
* Active COVID-19 infection
* Any history of underlying liver disorder, including hepatitis (see below)
* Any evidence of acute or chronic hepatitis B or C on screening testing
* Elevation of any or all liver enzymes (ALT, AST, total bilirubin) above the upper limit of normal (ULN) at baseline testing prior to enrollment
* A family history of hepatitis or currently living with a person who has been given a diagnosis of hepatitis
* A history of or currently working as a sex worker
* A history of or currently using intravenous (IV) drugs
* A self-reported history of alcoholic dependency or abuse
* A history of or current diagnosis of cardiovascular disease including heart failure, coronary artery disease, uncontrolled hypertension, uncontrolled diabetes; arrhythmias (or history of), or clinically relevant ECG abnormalities at baseline

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Osanetant on the testosterone levels. | 28 days
  We will test the ability of Osanetant to suppress testosterone production. A single arm pilot study of Osanetant at 200mg twice daily will be performed. Testosterone levels at baseline will be compared to levels at day 2, 3, 7 ,14, and 28 days of therapy. The overall effect of Osanetant on testosterone levels and the proportion of men achieving castrate levels of testosterone (<50ng/ml) will be assessed. Additionally, the reversibility of this effect will be assessed by evaluating the testosterone levels at 6-8 weeks posttreatment.

SECONDARY OUTCOMES:
To evaluate the effect of Osanetant on LH levels. | 28 days
  Levels of luteinizing hormone (LH) will be measured at baseline and days 2, 3, 7 ,14, and 28. These will be compared at each time point in order to assess the impact of NK3RA on these hormonal parameters.
To evaluate the effect of Osanetant on FSH levels. | 28 days
  Levels of follicle stimulating hormone (FSH) will be measured at baseline and days 2, 3, 7 ,14, and 28. These will be compared at each time point in order to assess the impact of NK3RA on these hormonal parameters.
To evaluate the effect of Osanetant on estradiol levels | 28 days
  Levels of estradiol will be measured at baseline and days 2, 3, 7 ,14, and 28. These will be compared at each time point in order to assess the impact of NK3RA on these hormonal parameters.
To evaluate the effect of Osanetant on PSA levels. | 28 days
  PSA will be compared at baseline and 28 days of therapy in order to evaluate the end biochemical efficacy of Osanetant on men with prostate cancer undergoing curative intent therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas, United States